CLINICAL TRIAL: NCT04240938
Title: Adult Encysted Dacryocystocele: Prevalence Among Patients With Epiphora and Its Management
Brief Title: Adult Dacryocystocele Among Patients With Epiphora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia2020
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lacrimal Passage Obstruction
MeSH Terms: interventions — Dacryocystorhinostomy

STUDY DESIGN:
Intervention Model Description: Adult Dacryocystocele
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lacrimal sac mucocele (Other): Adult patients with lacrimal sac mucocele
  Interventions: Procedure: Dacryocystorhinostomy

INTERVENTIONS:
Procedure: Dacryocystorhinostomy — Anastomosis between lacrimal sac and nasal cavity

SUMMARY:
Patients with lacrimal dacryocystocele were chosen for the study. Dacryocystorhinostomy were done for them after their evaluation.

DETAILED DESCRIPTION:
Evaluation for lacrimal passage in the included patients using syringing, probing and dye disappearance test. Dacryocystorhinostomy were done for all patients and followed up for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Lacrimal sac mucocele
* Acquired type

Exclusion Criteria:

* No previous lacrimal sac surgery
* Suspected lacrimal sac malignancy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Patency of the lacrimal passage | 2 weeks
  Disappearance of the watering of the eye reported by the patients and by fluorescein disappearance test
Disappearance of lacrimal sac swelling | 1 month
  No evident swelling in the medial side of the eye

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Ibrahiem, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No